CLINICAL TRIAL: NCT06780787
Title: Phase II Clinical Trial of FOLFOX, Botensilimab, Plus Balstilimab in Patients With Localized Rectal Cancer
Brief Title: FOLFOX, Botensilimab, and Balstilimab for the Treatment of Localized Rectal Cancer Before Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24589; NCI-2025-00072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24589 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rectal Adenocarcinoma; Stage IIA Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — balstilimab; Specimen Handling; Capecitabine; Endoscopic Mucosal Resection; Endoscopy; Biopsy; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin; Radiotherapy; Radiation; Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FOLFOX, botensilimab, balstilimab) (Experimental): Patients receive leucovorin calcium IV over 2 hours, oxaliplatin IV over 2 hours, and fluorouracil IV over 46 hours on day 1 of each cycle. Patients also receive botensilimab IV over 60 minutes on day 1 of cycles 1 and 4 and balstilimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients with complete clinical response may continue to receive balstilimab alone for an additional 12 cycles. Patients without complete clinical response may receive radiation therapy QD on weekdays and capecitabine PO BID concurrently on days of radiation therapy per standard of care. Additionally, patients undergo blood sample collection, biopsy with endoscopy exam, sigmoidoscopy, digital rectal exam, CT and MRI throughout the study.
  Interventions: Biological: Balstilimab; Procedure: Biospecimen Collection; Biological: Botensilimab; Drug: Capecitabine; Procedure: Computed Tomography; Procedure: Digital Rectal Examination; Procedure: Endoscopic Biopsy; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Radiation: Radiation Therapy; Procedure: Sigmoidoscopy

INTERVENTIONS:
Biological: Balstilimab — Given IV
  Other Names: AGEN 2034; AGEN-2034; AGEN2034
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Botensilimab — Given IV
  Other Names: AGEN 1181; AGEN-1181; AGEN1181; Anti-CTLA-4 Monoclonal Antibody AGEN1181
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Digital Rectal Examination — Undergo digital rectal exam
  Other Names: DRE
Procedure: Endoscopic Biopsy — Undergo biopsy with endoscopic exam
  Other Names: Endoscopy and Biopsy
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Sigmoidoscopy — Undergo sigmoidoscopy
  Other Names: Proctosigmoidoscopy

SUMMARY:
This phase II trial tests how well fluorouracil, oxaliplatin and leucovorin calcium (folinic acid) (FOLFOX) with botensilimab and balstilimab given before surgery (neoadjuvant) works in treating patients with rectal adenocarcinoma that has not spread to other parts of the body (localized). Currently, neoadjuvant therapy for rectal cancer includes chemotherapy and chemoradiation. Despite these aggressive treatments, only about half of patients achieve a complete clinical response. In fact, over half of rectal cancer patients go on to have surgery and often suffer post-surgery complications involving urine and bowel problems. Thus, there has been an increased focus on non-surgical treatments. Chemotherapy drugs, such as fluorouracil, oxaliplatin and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as botensilimab and balstilimab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving neoadjuvant FOLFOX with botensilimab and balstilimab may improve the rate of complete response and decrease the need for surgery and radiation therapy in patients with localized rectal adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the complete clinical response rate for patients with localized rectal cancer treated with neoadjuvant FOLFOX + botensilimab + balstilimab (FOLFOX-BB).

SECONDARY OBJECTIVES:

I. To evaluate the safety of FOLFOX-BB in patients with localized rectal cancer treated with neoadjuvant FOLFOX + botensilimab + balstilimab (FOLFOX-BB).

II. To estimate 3 year disease free survival rates in patients treated with FOLFOX-BB.

III. To estimate 3 year pelvic recurrence rates in patients with localized rectal cancer treated with neoadjuvant FOLFOX + botensilimab + balstilimab (FOLFOX-BB).

IV. To estimate the duration of response in patients with localized rectal cancer treated with neoadjuvant FOLFOX + botensilimab + balstilimab (FOLFOX-BB).

V. To evaluate 5 year survival rates in patients in patients with localized rectal cancer treated with neoadjuvant FOLFOX + botensilimab + balstilimab (FOLFOX-BB).

EXPLORATORY OBJECTIVES:

I. To examine changes in tumor microenvironment in response to FOLFOX-BB. II. To assess serial blood biomarkers to identify potential correlations with treatment response and outcomes.

OUTLINE:

Patients receive leucovorin calcium intravenously (IV) over 2 hours, oxaliplatin IV over 2 hours, and fluorouracil IV over 46 hours on day 1 of each cycle. Patients also receive botensilimab IV over 60 minutes on day 1 of cycles 1 and 4 and balstilimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients with complete clinical response may continue to receive balstilimab alone for an additional 12 cycles. Patients without complete clinical response may receive radiation therapy once daily (QD) on weekdays and capecitabine orally (PO) twice daily (BID) concurrently on days of radiation therapy per standard of care. Additionally, patients undergo blood sample collection, biopsy with endoscopy examination (exam), sigmoidoscopy, digital rectal exam, computed tomography (CT) and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patient are followed at 30 and 90 days, then every 3 months within 1 year of start of treatment, followed by every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Histologically confirmed adenocarcinoma of the rectum
* Rectal involvement defined as involvement of the rectum within 12 cm proximal from anal verge
* Radial margin of at least 3mm from the mesorectal fascia, with no threatened circumferential tumor margin based on MRI. No more than 4 lymph nodes (LN) with short axis > 1 cm
* T3N0, or TxN1 or TxN2 clinical stage based on MRI staging
* No evidence of distant metastatic disease based on imaging studies including CT chest and CT or MRI of abdomen and pelvis
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Without bone marrow involvement: Platelets ≥ 100,000/mm^3
* Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN
* Creatinine < 1.5 x ULN or clearance of ≥ 40 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 9 months for women, and at least 6 months for men, after the last dose of oxaliplatin therapy. If patients discontinue oxaliplatin more than 9 months (females) or 6 months (males) before discontinuation of balstilimab and/or botensilimab, females and males of childbearing potential must use an effective method of birth control or abstain from sexual activity for the course of the study through at least 120 days after the last dose of balstilimab and/or botensilimab

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Any treatment for rectal cancer prior to enrollment that includes (but not limited to) chemotherapy, radiation, and/or biological therapy
* Any prior immunotherapy
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Prior allogeneic organ transplantation
* Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement or biopsies
* Concurrent malignancy other than the diagnosis of rectal cancer, with the exception of curatively resected non-melanoma skin cancer, cervical cancer in situ, prostate cancer Gleason 6 or below that is localized to the prostate, or any other curatively resected cancer from which the patient remains in remission for at least 2 years without treatment
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation
* Clinically significant uncontrolled illness
* Females only: Pregnant or breastfeeding
* Prior allergic reaction or hypersensitivity to any of the study drug components
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs (excluding hypothyroidism, vitiligo, and psoriasis that is controlled with topical management)
* History of acute thrombotic venous events in the last 30 days before enrollment. If within 30 days, the patient should be on anticoagulants and without symptoms
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* History or current evidence of any condition, co-morbidity, therapy, any active infections (requiring antibiotics), or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Known previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to cycle 1 day 1 (C1D1)
* Uncontrolled infection with human immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV deoxyribonucleic acid (DNA) for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required
* Grade 2 or above neuropathy at the time of enrollment
* Dependence on total parenteral nutrition or intravenous hydration
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-11-05 (Estimated); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response (cCR) rate | At 3 months after treatment
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. Univariate logistic regression was used to estimate odds ratios (OR) and 90% confidence interval (CI) for cCR

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years
  ORR is calculated as the number of patients with complete response (per Response Evaluation Criteria in Solid Tumors version [v] 1.1) divided by the total number of treated/evaluable subjects. Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. Univariate logistic regression was used to estimate OR and 90% CI. Cox proportional hazards models were used to estimate hazard ratios (HR) with 95% CI.
Incidence of adverse events (AE) and serious adverse events (SAE) | Up to 90 days post-treatment
  AE and SAE will be described and graded at all dose levels using Common Terminology Criteria in Adverse Events v 5.0. Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables.
Disease free survival (DFS) | From the date of study enrollment until the recurrence of disease or death, whichever occurs first, assessed at 3 years post-treatment
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. Univariate logistic regression was used to estimate OR and 90% CI. Cox proportional hazards models were used to estimate HR with 95% CI. DFS distributions will be estimated using the Kaplan-Meier method.
Progression-free survival (PFS) | From the date of study enrollment until objective tumor progression or death, assessed up to 5 years
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. PFS distributions will be estimated using the Kaplan-Meier method. Kaplan-Meier method was used to plot PFS curves, and the log-rank test was applied to compare the distribution between groups. Cox proportional hazards models were used to estimate HR with 95% CI.
Pelvic recurrence rate | At 3 years after treatment
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables.
Duration of response (DOR) | From treatment response to progression or death, assessed up to 3 years
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. DOR distributions will be estimated using the Kaplan-Meier method.
Overall survival (OS) | From the date of study enrollment to the date of death, assessed up to 5 years post-treatment
  Data will be summarized using descriptive statistics for continuous variables and frequencies and percentages will be used for categorical variables. OS distributions will be estimated using the Kaplan-Meier method. Kaplan-Meier method was used to plot OS curves, and the log-rank test was applied to compare the distribution between groups. Cox proportional hazards models were used to estimate HR with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States